CLINICAL TRIAL: NCT03451513
Title: A Brief, Peer Co-led, Group-based Eating Disorder Prevention Program for Sexual Minority Young Adult Men
Brief Title: The Pride Body Project
Acronym: PBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Aaron Blashill, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HS-2017-0188; 1R01MD012698-01 (NIH)
Record Dates: First submitted 2018-02-20; First posted 2018-03-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Eating Disorder; Body Image
Keywords: Prevention; Sexual minority men; Internalization of the appearance ideal; Body dissatisfaction
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: On a phone screen, participants will be orally consented, and assessed briefly for eligibility. Participants who seem eligible will come in for an assessment made up of self- and clinician-report assessments, where they will be consented and assessed for eligibility. Eligible participants will be randomized. All participants completed intervention as determined by randomized assignment (i.e., MA or PBP). Each subject ID is pre-assigned to a study condition, determined by an online randomization program, prior to recruitment. Each eligible participant had a 1/2 chance to be assigned to either of the two study conditions. Participants will take part in two intervention sessions spaced a week apart. 1 to 2 weeks after the last session, participants will complete a follow-up, where they will do self- and clinician-report assessments. Further follow-up assessments, also comprised of both self- and clinician report assessments will be completed 6, 12, 18, and 24 months after treatment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator will not be told which condition individual participants are in. Outcome assessors at follow-up will not be told which condition the participant was in; any assessments regarding the content of intervention will be done by a separate, unblind assessor. The research assistants who enter the data from the clinician-based assessments administered by the outcome assessors will also be blind to participant condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pride Body Project (PBP) (Experimental): Participants assigned to this condition take part in a two-session intervention based on dissonance theory which encourages them to challenge the body ideal.
  Interventions: Behavioral: Pride Body Project
- Media Advocacy (MA) (Active Comparator): Participants assigned to this condition take place in a time and attention-matched active control where they discuss the role of media in promoting the body ideal.
  Interventions: Behavioral: Media Advocacy

INTERVENTIONS:
Behavioral: Pride Body Project — PBP is a 2-session eating disorder prevention program. Each session is 2 hours, and separated by a week. Groups have 4 to 7 participants and are led by a peer and a clinician. This program allows a forum for young men to critique the appearance ideal. These exercises should induce cognitive dissonance, which subsequently lead to a reduction of internalization of the ideal. In session 1, participants: (1) define the "ideal" body type in the gay community, (2) discuss its origin and perpetration, (3) brainstorm its costs, (4) participate in a verbal challenge where they counter the "ideal," and (5) are asked to complete three assignments. In session 2, participants: (1) review homework, (2) engage in role-plays to counter pursuit of the "ideal," (3) discuss ways to challenge "body talk" statements, (4) list ways to resist the pressure to pursue this "ideal" (body activism), (5) discuss barriers to body activism and how to overcome those barriers, and (6) select an exit activity.
  Arms: Pride Body Project (PBP)
Behavioral: Media Advocacy — We will use a media advocacy (MA) intervention as an active, time- and attention-matched control. MA is a 2 session, group-based program with co-leaders (1 peer and 1 clinician). The MA content centers on acknowledging and discussing the role the media has on shaping body image ideals. In session 1, there is a discussion on describing the ideal body in the gay community and how the media impacts this ideal. Following this, participants will watch a video on how the media influences body image among gay men, and the consequences of internalizing these messages. In session 2, participants will watch a second video. Next, the group discusses other forms of media (e.g., pornography, social media) and how it impacts body image.
  Arms: Media Advocacy (MA)

SUMMARY:
The purpose of this study is to better investigate the efficacy of the PRIDE Body Project in respect to preventing eating disorders in sexual minority men. In this randomized controlled trial, participants will be enrolled in one of two arms: 1) the PRIDE Body Project intervention or 2) Media Advocacy, a time and attention-matched intervention. This study will recruit participants who are between the ages of 18 and 35, identify as men, are gay, bisexual, or experience sexual attraction to men, and who express body image concerns for the San Diego area.

DETAILED DESCRIPTION:
Eating disorders (i.e., anorexia nervosa, bulimia nervosa, binge eating disorder, and eating disorder not otherwise specified) are resistant to treatment and associated with significant morbidity and mortality. Thus, efficacious and efficient eating disorder prevention programs are greatly needed. Extant literature has found that males also experience eating disorders, constituting up to 40% of individuals with diagnostic/sub-threshold eating pathology.

Among males, sexual minorities (i.e., gay, bisexual, and non-heterosexual identified individuals) are a salient subgroup that is at substantial risk for developing eating disorders. Indeed, sexual minority males are not only at elevated risk compared to heterosexual males, but are also at elevated risk compared to heterosexual females. The lifetime prevalence for any eating disorder diagnosis among sexual minority males is 8.8%, and subclinical diagnosis is 15.6%. This is in contrast to heterosexual females, in which the prevalence for clinical and subclinical diagnoses are at 4.8% and 8.0%, respectively. These findings indicate that sexual minority males are one of the most vulnerable groups in regard to eating pathology risk.

Despite their high vulnerability, there is a paucity of research on eating disorder prevention programs among sexual minority males. The investigators are only aware of one previous prevention program targeting sexual minority males. The PRIDE Body Project, developed and tested by this research team, is a two-session, peer co-led, group, cognitive dissonance-based eating disorder prevention program, based on existing eating disorder prevention programs developed with females (The Body Project). In the preliminary randomized controlled trial (RCT), the researchers found significant and large effects on eating pathology and relevant eating disorder risk factors, compared to a waitlist control condition, at post-treatment and 4-weeks post-treatment. Additionally, preliminary mediation analyses revealed that internalization of the appearance ideal and body dissatisfaction accounted for significant variance in the relationship between treatment condition and eating pathology. These results represent an important first step in demonstrating the acceptability, feasibility, and preliminary efficacy of a brief, peer-led eating disorder prevention program for sexual minority males.

Despite these initial findings, future research is needed to further test this promising intervention. Specifically, it is not known if the PRIDE Body Project will exert a clinically and statistically significant effect in comparison to a time and attention-matched control condition. Additionally, it is unknown if the intervention effects will persist beyond 4-weeks post-intervention. To address these gaps, we propose the following aims:

Specific Aim 1: Conduct a randomized controlled trial assessing the PRIDE Body Project to a time and attention-matched active control condition. The researchers plan to randomize 348 18 to 35-year-old sexual minority males (in a 1:1 scheme) to either the experimental PRIDE Body Project condition or a media advocacy condition. Participants will be followed for 2 years post-baseline assessment, with major assessment points at: baseline, post-intervention, 6 month, 12 month, 18 month, and 24 month follow-up. Primary outcomes will be eating disorder symptoms and eating disorder onset. The researchers hypothesize that participants randomized to the PRIDE Body Project will yield significantly greater reductions in eating disorder symptoms, and produce lower incidence rates of eating disorders, compared to participants in the media advocacy condition.

Specific Aim 2: Conduct longitudinal mediation analyses of the treatment effect. In an effort to more fully understand the mechanisms of change in the PRIDE Body Project, the researchers will assess two theoretically and empirically based mediators of the effect of treatment on eating disorder symptoms. Specifically, the researchers hypothesize that assignment to the PRIDE Body Project condition will lead to significant reductions in body dissatisfaction and internalization of the appearance ideal, which in turn will lead to reductions in eating disorder symptoms/onset.

Sexual minority males are one of the most vulnerable groups for developing eating disorders, yet the creation and testing of theoretically and empirically based prevention programs is in its very early stages. The proposed study will provide crucial information on the efficacy of a promising eating disorder prevention program, and has the potential to impact this vulnerable population of young males. Given the brevity of the program, and its emphasis on peer co-leaders, it has high potential for implementation and public health impact. This proposal is also aligned with the purpose and research priorities of PA-15-261 (The Health of Sexual and Gender Minority (SGM) Populations), namely, interventions aimed to "ameliorate health disparities in SGM" through "large-scale design, implementation and evaluation of preventative and/or treatment interventions addressing health issues in SGM populations."

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35
* Male gender
* Identifies as gay or bisexual or reports sexual attraction to men
* Reports body image concerns
* Able to provide informed consent

Exclusion Criteria:

* Diagnosis of an eating disorder (anorexia nervosa, bulimia nervosa, binge eating disorder)
* Significant neuropsychiatric illness (e.g., diagnosis of dementia, untreated bipolar disorder, psychosis, or active suicidal ideation)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In order to be eligible, participants must identify as men.
Enrollment: 453 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination, Edition 17.0 (EDE-17) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Assess changes in eating disorder symptoms and diagnosis
Eating Pathology Symptoms Inventory | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Assess changes in pathological eating behaviors

SECONDARY OUTCOMES:
Sociocultural Attitudes Towards Appearance Questionnaire 3 (SATAQ-3) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Assess internalization of appearance ideal and societal pressure to achieve that ideal
Sociocultural Attitudes Towards Appearance Questionnaire Revised (SATAQ-4R) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Assess internalization of appearance ideal and societal pressure to achieve that ideal
Male Body Attitudes Scale/Revised (MBAS-R) | Baseline assessment; 1 to 2 week post-intervention assessment, 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report measure assessing muscle, fat, and height dissatisfaction
Depression, Anxiety, Stress Scale (DASS) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Measures symptoms of depression, anxiety, and stress (non-specific physiological arousal), all contribute to psychological distress (i.e., negative affect)
Drive for Muscularity Scale (DMS) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report measure of muscularity-oriented body image and behaviors
Self-Objectification Scale (SOQ) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Assess degree to which participant sees their body in an objectified, appearance-based manner v. a non-objectified, competence-based manner
Partner Objectification Scale (POS) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  10 items based on the SOQ which assess degree to which participant sees the bodies of potential partners in an objectified, appearance-based manner v. a non-objectified, competence-based manner
Steroid and Appearance Related Drug Items (APEDS) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Item assess frequency of use of seven drugs that are classified as steroids or are used to change appearance
Sexual Risk Behaviors (SRB) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  5 item questionnaire assessing frequency of risky sexual behavior (unprotected sex with partners of unknown HIV status), as well as PrEP use
Dysmorphic Concerns Questionnaire (DCQ) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report measure of body dysmorphic disorder symptoms
Muscle Dysmorphic Disorder Inventory (MDDI) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report measure of body dysmorphic disorder symptoms
MINI-International Neuropsychiatric Interview MINI | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Clinician-based interview for psychiatric disorders
NIDA-CTN Addictions Severity Index Lite (ASI-Lite) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Clinician-based interview for substance and alcohol use
BMI Calculations | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Measurement of height and weight
Gender Identity Questionnaire (Gender Identity) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report based measure of gender identity
The Coronavirus Health Impact Survey (Crisis) V0.2 Adult Self-report Baseline Form | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report based measure to assess the effects of COVID-19 on daily functions and mental health
United States Department of Agriculture (USDA) Food and Nutrition Services US Household Food Security Survey Module | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report based measure for food insecurity
Importance of Gay/Bisexual Community Activities (IBGCA) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report based measure for community involvement
Structured Clinical Interview for DSM-IV-TR Body Dysmorphic Module (SCID BDD Module) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Clinician-based interview for Body Dysmorphic Disorder
Social Justice Sexuality Survey (SJSS) | Baseline assessment; 1 to 2 week post-intervention assessment; 6 month follow-up assessment; 12 month follow-up assessment; 18 month follow-up assessment; 24 month follow-up assessment
  Self-report based measure for community involvement

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Blashill, Ph.D., Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klump KL, Bulik CM, Kaye WH, Treasure J, Tyson E. Academy for eating disorders position paper: eating disorders are serious mental illnesses. Int J Eat Disord. 2009 Mar;42(2):97-103. doi: 10.1002/eat.20589. No abstract available. PMID 18951455
- [Background] Mitchell JE, Crow S. Medical complications of anorexia nervosa and bulimia nervosa. Curr Opin Psychiatry. 2006 Jul;19(4):438-43. doi: 10.1097/01.yco.0000228768.79097.3e. PMID 16721178
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- [Background] Brownley KA, Berkman ND, Sedway JA, Lohr KN, Bulik CM. Binge eating disorder treatment: a systematic review of randomized controlled trials. Int J Eat Disord. 2007 May;40(4):337-48. doi: 10.1002/eat.20370. PMID 17370289
- [Background] Hudson JI, Hiripi E, Pope HG Jr, Kessler RC. The prevalence and correlates of eating disorders in the National Comorbidity Survey Replication. Biol Psychiatry. 2007 Feb 1;61(3):348-58. doi: 10.1016/j.biopsych.2006.03.040. Epub 2006 Jul 3. PMID 16815322
- [Background] Russell CJ, Keel PK. Homosexuality as a specific risk factor for eating disorders in men. Int J Eat Disord. 2002 Apr;31(3):300-6. doi: 10.1002/eat.10036. PMID 11920991
- [Background] Brown TA, Keel PK. The impact of relationships, friendships, and work on the association between sexual orientation and disordered eating in men. Eat Disord. 2013;21(4):342-59. doi: 10.1080/10640266.2013.797825. PMID 23767674
- [Background] Feldman MB, Meyer IH. Eating disorders in diverse lesbian, gay, and bisexual populations. Int J Eat Disord. 2007 Apr;40(3):218-26. doi: 10.1002/eat.20360. PMID 17262818
- [Background] Brown TA, Keel PK. A randomized controlled trial of a peer co-led dissonance-based eating disorder prevention program for gay men. Behav Res Ther. 2015 Nov;74:1-10. doi: 10.1016/j.brat.2015.08.008. Epub 2015 Sep 3. PMID 26342904
- [Background] Stice E, Marti CN, Spoor S, Presnell K, Shaw H. Dissonance and healthy weight eating disorder prevention programs: long-term effects from a randomized efficacy trial. J Consult Clin Psychol. 2008 Apr;76(2):329-40. doi: 10.1037/0022-006X.76.2.329. PMID 18377128
- [Background] Stice E, Rohde P, Gau J, Shaw H. An effectiveness trial of a dissonance-based eating disorder prevention program for high-risk adolescent girls. J Consult Clin Psychol. 2009 Oct;77(5):825-34. doi: 10.1037/a0016132. PMID 19803563
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871